CLINICAL TRIAL: NCT06205082
Title: A Multicenter, Open Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of LIT-00814 Tablets in Patients With Advanced Solid Tumor/Esophageal Cancer.
Brief Title: A Phase I Clinical Trial to Evaluate LIT-00814 Tablets in Patients With Advanced Solid Tumor
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: LittDD Medicines Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIT-00814-2023-CP101
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LIT-00814 20mg (Experimental): Take a fixed dose of LIT-00814 tablets orally once a day in the morning and evening, and take them orally continuously.
  Interventions: Drug: LIT-00814
- LIT-00814 50mg (Experimental): Take a fixed dose of LIT-00814 tablets orally once a day in the morning and evening, and take them orally continuously.
  Interventions: Drug: LIT-00814
- LIT-00814 100mg (Experimental): Take a fixed dose of LIT-00814 tablets orally once a day in the morning and evening, and take them orally continuously.
  Interventions: Drug: LIT-00814
- LIT-00814 150mg (Experimental): Take a fixed dose of LIT-00814 tablets orally once a day in the morning and evening, and take them orally continuously.
  Interventions: Drug: LIT-00814

INTERVENTIONS:
Drug: LIT-00814 — LIT-00814 is an oral tablet.

SUMMARY:
This study is a multi-center, open, dose-increasing and dose-expanding phase I clinical study, aiming at evaluating the safety, tolerability, pharmacokinetic characteristics and preliminary anti-tumor activity of LIT-00814 tablets with different doses in China, and preliminarily evaluating the relationship between biomarkers and anti-tumor activity of LIT-00814 tablets.

This study includes two parts: Ia phase (i.e. dose escalation) and Ib phase (i.e. dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal representative shall voluntarily sign the informed consent approved by the Ethics Committee before starting any screening procedure.
2. Male or female, age ≥18 years old.
3. Unresectable locally advanced or metastatic solid tumor confirmed by histology or cytology.
4. Subjects with relapsed and/or metastatic advanced solid tumors who have failed or have no standard treatment at present, or who are unable to accept standard treatment.
5. At least one target lesion.
6. ECOG score 0~1.
7. Subjects must have sufficient organ function.
8. Agree to use effective contraceptive measures within 3 months (about 90 days) from the signing of informed consent to the last administration of the study drug.

Exclusion Criteria:

1. The toxicity caused by previous treatment did not recover to ≤1 grade before the first study administration;
2. Known or symptomatic active central nervous system (CNS) metastasis or cancerous meningitis in the screening period;
3. Patients who have undergone surgery within 28 days before the first administration and have not recovered yet;
4. Suffering from uncontrolled or clinically significant cardiovascular diseases;
5. Other malignant tumors occurred within 3 years before the first administration;
6. Patients with active chronic hepatitis B, or patients with active hepatitis C, or patients with human immunodeficiency virus (HIV-Ab positive) or syphilis infection;
7. There are circumstances that affect the subjects' compliance with the research plan;
8. Other circumstances that the researcher thinks are not suitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-10-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days post last drug administration
Determination of the MTD and RP2D of LIT-00814 monotherapy | 24 days after the first dose
  Defined as the highest dose level at which no more than 1 of 6 subjects experience a DLT during the DLT assessment window（24days）

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Until documented the disease progresses or informed consent is withdrawn
  according to the criterion of RECIST1.1, the proportion of subjects with complete remission (CR) and partial remission (PR) during the study period.
Disease control rate (DCR) | Until documented the disease progresses or informed consent is withdrawn
  According to the criterion of RECIST1.1, the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) during the study period.
Disease progression-free survival (PFS) | Until documented the disease progresses or informed consent is withdrawn
  It is defined as the time between the first administration date of the study drug and the disease progression or death, whichever occurs first.
Treatment onset time (TTR) | Until documented the disease progresses or informed consent is withdrawn
  It is defined as the time between the first administration date of the study drug and the first determination of complete remission (CR) and partial remission (PR).
Overall survival (OS) | date of death from any cause or withdrawal of informed consent
  The time from the first administration date of the study drug to the death (for any reason) of the subject.
Pharmacokinetic parameters：Maximum observed concentration（Cmax） | C0D1-D3 0-72h（single dose），C1D1 0h、C1D8 0h、C2D1 0-8h（21days/cycle）
  Maximum concentration of LIT-00814 in blood after single dose and continuous multiple doses
Pharmacokinetic parameters：Area under the concentration-time curve (AUC) | C0D1-D3 0-72h（single dose），C1D1 0h、C1D8 0h、C2D1 0-8h（21days/cycle）
  The concentration of LIT-00814 in blood after single dose and continuous multiple doses
Pharmacokinetic parameters：Half-life (t1/2) | C0D1-D3 0-72h（single dose），C1D1 0h、C1D8 0h、C2D1 0-8h（21days/cycle）
  The concentration of LIT-00814 in blood after single dose and continuous multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China